CLINICAL TRIAL: NCT03664128
Title: Pregnancy and Anxious Thoughts: The Role of the Immune and Endocrine Systems
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Brain & Behavior Research Foundation (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00087653; 1K23MH110607-01A1 (NIH)
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-06

CONDITIONS: Perinatal Anxiety
MeSH Terms: interventions — Coping Skills; Pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants' blood will be drawn (up to 55 ml) at all four sessions by a study clinician or a trained research assistant. Blood will be collected in sodium-heparin tubes for immune cell preparation. Peripheral blood mononuclear cell (PBMC) suspensions will be prepared within 8 hours of blood collection by low-density gradient centrifugation via a Hermle Z 300 K #55085010, to avoid erythrophagy-related activation of the monocytes. PBMCs will be frozen and stored at -80° C using 10% dimethylsulfoxide, thereby allowing all samples to be analyzed in parallel.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pregnant women positive for anxiety: 100 pregnant women who screen positive for anxiety symptoms (>21 on the Perinatal Anxiety Screening Scale). Participants are matched for age, parity, and gestational age at enrollment.
  Coping with Anxiety through Living Mindfully (CALM) Pregnancy: Mindfulness-based Cognitive Behavioral Therapy (CBT) for perinatal anxiety on a subset (8 participants)
  Interventions: Other: Coping with Anxiety through Living Mindfully (CALM) Pregnancy
- healthy pregnant controls: 100 matched healthy pregnant women. Participants are matched for age, parity, and gestational age at enrollment.

INTERVENTIONS:
Other: Coping with Anxiety through Living Mindfully (CALM) Pregnancy — Mindfulness-based Cognitive Behavioral Therapy (CBT) for perinatal anxiety on a subset (8 participants); no intervention for other participants
  Groups: pregnant women positive for anxiety

SUMMARY:
The aim of the proposed research is to identify the clinical and biological phenotypes that define perinatal anxiety. The importance of this research to public health is that it will help to identify women at high risk, and will also serve as the basis for further studies that would identify genetic and epigenetic markers of risk and lead to research to identify novel treatment targets. The research is based upon preliminary data demonstrating a relationship between inflammatory cytokines and Trait anxiety in pregnancy; between progesterone and postpartum anxiety; and between allopregnanolone and obsessive symptoms in pregnancy. The proposed research will build upon these preliminary findings by prospectively examining the clinical features of anxiety in a cohort of pregnant women and healthy matched controls, and by analyzing blood samples from the same cohort for inflammatory cytokines, reproductive hormones, and immune cell types. The proposed study will therefore identify the clinical and biological phenotypes that characterize perinatal anxiety and will identify potential novel targets for treatment.

DETAILED DESCRIPTION:
My preliminary data from the Viral Immunity in Pregnancy Study found a strong association in 49 pregnant women between levels of anxiety and of cytokines. When the investigators controlled for clinical confounders, some of those associations disappeared - but there was still a strong correlation between anxiety score and the cytokine interleukin (IL) 6.

Hypothesis: Anxious pregnant women (as determined by a score > 21 on the Perinatal Anxiety Screening Scale (PASS)) will have elevated pro-inflammatory cytokines in pregnancy (at second and third trimesters) and will demonstrate greater continued elevation at 6 weeks and 6 months postpartum when compared to healthy controls. Leukocyte subpopulation analysis in anxious women will show a higher ratio of T-helper 1-type (Th1) to T-helper 2- type (Th2) cells and a greater monocyte activation across the perinatal period than that in healthy controls.

Hypothesis: There will be a negative correlation between allopregnanolone (ALLO) and pro-inflammatory markers (as listed above in primary outcome measure) in pregnancy, and between allopregnanolone (ALLO) in pregnancy and pro-inflammatory markers in the postpartum.

Hypothesis: Women with a pro-inflammatory immune fingerprint and low levels of allopregnanolone (ALLO) as determined by outcomes 1 and 2 will show increased attentional bias to threat, as demonstrated by measurement of autonomic reactivity in response to a validated pregnancy-specific modified Stroop task.

Hypothesis: Anxious pregnant women will find it feasible and acceptable to engage in a mindfulness-based cognitive behavioral therapy intervention for perinatal anxiety.

For each of these, the investigators will compare the outcome between anxious and non-anxious women.

The current study has 2 parts. The initial part, funded by Brain and Behavior Foundation, was designed to collect general information about the immune and endocrine mechanisms of perinatal anxiety and to test following aims:

Aim 1: To determine if obsessional anxiety in pregnancy corresponds to changes in immune functioning.

Aim 2: To determine if symptoms of obsessional anxiety in pregnancy are associated with changes in the levels of progesterone and its metabolites.

Aim 3: To determine feasibility and acceptability of mindfulness-based cognitive behavioral intervention designed to ameliorate prenatal anxiety and the accompanying inflammatory dysregulation.

I next expanded the study to obtain more detailed biological data; There is no intervention in the expansion for this phase.

I plan to recruit a group of 200 pregnant women (100 who screen positive for anxiety and 100 healthy controls). Subjects will answer questionnaires about mood and anxiety symptoms and have participants' blood drawn at four visits across pregnancy and the postpartum; in the second visit, participants will also perform a computer task designed to test how well participants can inhibit responses. A small subset of subjects will enroll in a group mindfulness intervention as well. This study is designed to achieve the following aims:

1. To compare the "immune fingerprint" of women with significant perinatal anxiety with that of a cohort of healthy matched controls.
2. To determine how perinatal changes in the "immune fingerprint" relate to changes in levels of progesterone metabolites (specifically, allopregnanolone) across pregnancy.
3. To identify how changes in the "immune fingerprint" and progesterone metabolites are related to changes in maternal response to threat.

This study is an effort to further characterize the role of the immune system in common psychiatric symptomatology and the likely bidirectional relationship between the immune system and reproductive hormones that may be related to disease flares among a subset of patients. This work could eventually extend to the gene signatures responsible for immune pathways, to epigenetic studies, and/or to brain imaging studies examining differences in brain region function as affected by inflammation. Ultimately, this would allow the investigators to augment the traditional psychopharmacological focus on serotonin modification with new treatment targets, including cytokines, intracellular inflammatory mediators, neurogenesis, or glial cell activation.

ELIGIBILITY:
Inclusion Criteria for all:

* Pregnant and <27 weeks gestation
* Age 18 or above
* Able to provide written consent
* Healthy pregnancy.

Additional inclusion criteria specific to anxiety group:

* Significant anxiety symptoms as measured by a score of > 21 on the Perinatal Anxiety Screening Scale (PASS)
* a diagnosis of current anxiety disorder by Structured Clinical Interview for Diagnostic And Statistical Manual Of Mental Disorders (DSM) V Diagnoses (SCID), or a diagnosis of a current anxiety disorder by a clinician interview using DSM-V criteria.

Exclusion Criteria for all:

* Multifetal pregnancy
* Autoimmune or endocrine disease
* Meeting criteria for a major depressive episode at study entry
* Active suicidal ideation at study entry
* Bipolar disorder or primary psychotic disorder
* Recent or current substance abuse.

Additional exclusion criteria for healthy controls:

* No history of an anxiety or depressive disorder as determined by Structured Clinical Interview for DSM-V Diagnoses (SCID)
* No current use of an antidepressant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant Women with or without mental health history.
Sampling Method: Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2016-06-24 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Changes in the level of interleukin 6 (IL-6) | 4 study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation; 3) 6 weeks postpartum; 4) 6 months postpartum
  The MesoScale Discovery Pro-Inflammatory Multiplex Assay will be used to measure concentrations of IL-6 in pg/mL. Concentration will be log-transformed.
Changes in the level of Interleukin 15 (IL-15) | 4 study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation; 3)6 weeks postpartum; 4) 6 months postpartum
  The MesoScale Discovery Pro-Inflammatory Multiplex Assay will be used to measure concentrations of IL-15 in pg/mL. Concentration will be log-transformed.
Changes in the level of Granulocyte macrophage colony stimulating factor (GM-CSF) | 4 study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation; 3)6 weeks postpartum; 4) 6 months postpartum
  The MesoScale Discovery Pro-Inflammatory Multiplex Assay will be used to measure concentrations of GM-CSF in pg/mL. Concentration will be log-transformed.
Changes in the level of Granulocyte colony stimulating factor (G-CSF) | 4 study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation; 3)6 weeks postpartum; 4) 6 months postpartum
  The MesoScale Discovery Pro-Inflammatory Multiplex Assay will be used to measure concentrations of G-CSF in pg/mL. Concentration will be log-transformed.
Changes in the level of Chemokine C-X-C motif ligand 8 (CXCL8) | 4 study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation; 3)6 weeks postpartum; 4) 6 months postpartum
  The MesoScale Discovery Pro-Inflammatory Multiplex Assay will be used to measure concentrations of C-X-CL8 in pg/mL. Concentration will be log-transformed.
Changes in the level of Chemokine C-C motif ligand 3 (CCL3) | 4 study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation; 3)6 weeks postpartum; 4) 6 months postpartum
  The MesoScale Discovery Pro-Inflammatory Multiplex Assay will be used to measure concentrations of CCL3 in pg/mL. Concentration will be log-transformed.
Leukocyte subpopulation | Second study visit (32-36 weeks gestation)
  The investigators will use flow cytometry and fluorescence activated cell-sorting analysis to determine the percentages of leukocyte subpopulations, namely T cells, B cells, natural killer cells, monocytes, macrophages, and dendritic cells.

SECONDARY OUTCOMES:
Relationship of changes in levels of allopregnanolone (ALLO) to pro-inflammatory markers | 1st and 2nd study visits: 1) 22-26 weeks gestation; 2) 32-36 weeks gestation
  The investigators will use enzyme-linked immunosorbent assay (ELISA) to measure levels of ALLO in ng/mL, across pregnancy and calculate the rate of change across pregnancy to determine if there is any correlation between the level of ALLO at second and third trimesters and levels of the pro-inflammatory markers listed above.
Heart Rate Variability | Second study visit (32-36 weeks gestation)
  The investigators will measure high-frequency heart rate variability (in length of R to R interval in milliseconds, using electrocardiogram in Biopac Data Acquisition System) at baseline and in response to a stressor. This will be analyzed to see if there is a change comparing women with elevated inflammation and decreased ALLO to those without these features.
Electrodermal Activity | Second study visit (32-36 weeks gestation)
  The investigators will measure electrodermal activity on the hands at baseline and in response to a stressor, using Biopac Data Acquisition System and electrodermal activity electrodes. The investigators will analyze these data to assess any changes when comparing women with elevated inflammation and decreased ALLO to those without these features.
Feasibility of a mindfulness-based cognitive behavioral therapy intervention as assessed by participant retention number | Study visit (22-36 weeks gestation)
  The investigators will measure feasibility of this intervention by enrollment and retention of participants in a mindfulness-based cognitive behavioral therapy intervention for perinatal anxiety (CALM pregnancy). The intervention will be deemed feasible if the investigators successfully enroll at least 6 participants, and all participants complete at least 6 of the 8 sessions.
Acceptability of a mindfulness-based cognitive behavioral therapy intervention as assessed by a Likert scale | Study visit (22-36 weeks gestation)
  The investigators will measure acceptability of the CALM pregnancy intervention to participants using a Likert scale (1-5, with 1 being not at all acceptable and 5 being very acceptable).

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Osborne, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Women's Mood Disorders Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alder J, Fink N, Bitzer J, Hosli I, Holzgreve W. Depression and anxiety during pregnancy: a risk factor for obstetric, fetal and neonatal outcome? A critical review of the literature. J Matern Fetal Neonatal Med. 2007 Mar;20(3):189-209. doi: 10.1080/14767050701209560. PMID 17437220
- [Background] Andersson L, Sundstrom-Poromaa I, Wulff M, Astrom M, Bixo M. Implications of antenatal depression and anxiety for obstetric outcome. Obstet Gynecol. 2004 Sep;104(3):467-76. doi: 10.1097/01.AOG.0000135277.04565.e9. PMID 15339755
- [Background] Ashley V, Honzel N, Larsen J, Justus T, Swick D. Attentional bias for trauma-related words: exaggerated emotional Stroop effect in Afghanistan and Iraq war veterans with PTSD. BMC Psychiatry. 2013 Mar 14;13:86. doi: 10.1186/1471-244X-13-86. PMID 23496805
- [Background] Bar-Shai M, Gott D, Kreinin I, Marmor S. Atypical presentations of pregnancy-specific generalized anxiety disorders in women without a previous psychiatric background. Psychosomatics. 2015 May-Jun;56(3):286-91. doi: 10.1016/j.psym.2013.12.017. Epub 2014 Jan 1. No abstract available. PMID 25262048
- [Background] Backstrom T, Bixo M, Johansson M, Nyberg S, Ossewaarde L, Ragagnin G, Savic I, Stromberg J, Timby E, van Broekhoven F, van Wingen G. Allopregnanolone and mood disorders. Prog Neurobiol. 2014 Feb;113:88-94. doi: 10.1016/j.pneurobio.2013.07.005. Epub 2013 Aug 23. PMID 23978486
- [Background] Baer AN, Witter FR, Petri M. Lupus and pregnancy. Obstet Gynecol Surv. 2011 Oct;66(10):639-53. doi: 10.1097/OGX.0b013e318239e1ee. PMID 22112525
- [Background] Bergink V, Burgerhout KM, Weigelt K, Pop VJ, de Wit H, Drexhage RC, Kushner SA, Drexhage HA. Immune system dysregulation in first-onset postpartum psychosis. Biol Psychiatry. 2013 May 15;73(10):1000-7. doi: 10.1016/j.biopsych.2012.11.006. Epub 2012 Dec 25. PMID 23270599
- [Background] Biggio G, Pisu MG, Biggio F, Serra M. Allopregnanolone modulation of HPA axis function in the adult rat. Psychopharmacology (Berl). 2014 Sep;231(17):3437-44. doi: 10.1007/s00213-014-3521-6. PMID 24658404
- [Background] Brunton PJ. Neuroactive steroids and stress axis regulation: Pregnancy and beyond. J Steroid Biochem Mol Biol. 2016 Jun;160:160-8. doi: 10.1016/j.jsbmb.2015.08.003. Epub 2015 Aug 7. PMID 26259885
- [Background] Buyon JP. The effects of pregnancy on autoimmune diseases. J Leukoc Biol. 1998 Mar;63(3):281-7. doi: 10.1002/jlb.63.3.281. PMID 9500514
- [Background] Chen SJ, Liu YL, Sytwu HK. Immunologic regulation in pregnancy: from mechanism to therapeutic strategy for immunomodulation. Clin Dev Immunol. 2012;2012:258391. doi: 10.1155/2012/258391. Epub 2011 Nov 3. PMID 22110530
- [Background] Coe CL. Maternal anxiety during pregnancy influences infant responses to immunization. Brain Behav Immun. 2013 Aug;32:19-20. doi: 10.1016/j.bbi.2013.05.004. Epub 2013 May 21. No abstract available. PMID 23707424
- [Background] Coussons-Read ME, Okun ML, Nettles CD. Psychosocial stress increases inflammatory markers and alters cytokine production across pregnancy. Brain Behav Immun. 2007 Mar;21(3):343-50. doi: 10.1016/j.bbi.2006.08.006. Epub 2006 Oct 6. PMID 17029703
- [Background] Dayan J, Creveuil C, Herlicoviez M, Herbel C, Baranger E, Savoye C, Thouin A. Role of anxiety and depression in the onset of spontaneous preterm labor. Am J Epidemiol. 2002 Feb 15;155(4):293-301. doi: 10.1093/aje/155.4.293. PMID 11836191
- [Background] 74 Diggle P, Heagerty P, Liang K-Y, and Zeger S. Analysis of Longitudinal Data. 2nd edition. Oxford Statistical Science Series: 25. Oxford: Oxford University Press, 2002.
- [Background] DiPietro JA, Costigan KA, Gurewitsch ED. Fetal response to induced maternal stress. Early Hum Dev. 2003 Nov;74(2):125-38. doi: 10.1016/j.earlhumdev.2003.07.001. PMID 14580752
- [Background] Duivis HE, Vogelzangs N, Kupper N, de Jonge P, Penninx BW. Differential association of somatic and cognitive symptoms of depression and anxiety with inflammation: findings from the Netherlands Study of Depression and Anxiety (NESDA). Psychoneuroendocrinology. 2013 Sep;38(9):1573-85. doi: 10.1016/j.psyneuen.2013.01.002. Epub 2013 Feb 8. PMID 23399050
- [Background] Dunkel Schetter C, Tanner L. Anxiety, depression and stress in pregnancy: implications for mothers, children, research, and practice. Curr Opin Psychiatry. 2012 Mar;25(2):141-8. doi: 10.1097/YCO.0b013e3283503680. PMID 22262028
- [Background] Field T, Diego M, Hernandez-Reif M, Schanberg S, Kuhn C, Yando R, Bendell D. Pregnancy anxiety and comorbid depression and anger: effects on the fetus and neonate. Depress Anxiety. 2003;17(3):140-51. doi: 10.1002/da.10071. PMID 12768648
- [Background] Field T. Prenatal depression effects on early development: a review. Infant Behav Dev. 2011 Feb;34(1):1-14. doi: 10.1016/j.infbeh.2010.09.008. PMID 20970195
- [Background] Furtado M, Katzman MA. Neuroinflammatory pathways in anxiety, posttraumatic stress, and obsessive compulsive disorders. Psychiatry Res. 2015 Sep 30;229(1-2):37-48. doi: 10.1016/j.psychres.2015.05.036. Epub 2015 Jun 6. PMID 26296951
- [Background] Gao J. Correlation between anxiety-depression status and cytokines in diarrhea-predominant irritable bowel syndrome. Exp Ther Med. 2013 Jul;6(1):93-96. doi: 10.3892/etm.2013.1101. Epub 2013 May 8. PMID 23935726
- [Background] Gilbert Evans SE, Ross LE, Sellers EM, Purdy RH, Romach MK. 3alpha-reduced neuroactive steroids and their precursors during pregnancy and the postpartum period. Gynecol Endocrinol. 2005 Nov;21(5):268-79. doi: 10.1080/09513590500361747. PMID 16373246
- [Background] Glover V. Maternal depression, anxiety and stress during pregnancy and child outcome; what needs to be done. Best Pract Res Clin Obstet Gynaecol. 2014 Jan;28(1):25-35. doi: 10.1016/j.bpobgyn.2013.08.017. Epub 2013 Sep 18. PMID 24090740
- [Background] Goodman JH, Guarino A, Chenausky K, Klein L, Prager J, Petersen R, Forget A, Freeman M. CALM Pregnancy: results of a pilot study of mindfulness-based cognitive therapy for perinatal anxiety. Arch Womens Ment Health. 2014 Oct;17(5):373-87. doi: 10.1007/s00737-013-0402-7. Epub 2014 Jan 22. PMID 24449191
- [Background] Grace SL, Evindar A, Stewart DE. The effect of postpartum depression on child cognitive development and behavior: a review and critical analysis of the literature. Arch Womens Ment Health. 2003 Nov;6(4):263-74. doi: 10.1007/s00737-003-0024-6. PMID 14628179
- [Background] Guintivano J, Arad M, Gould TD, Payne JL, Kaminsky ZA. Antenatal prediction of postpartum depression with blood DNA methylation biomarkers. Mol Psychiatry. 2014 May;19(5):560-7. doi: 10.1038/mp.2013.62. Epub 2013 May 21. PMID 23689534
- [Background] Haupl T, Ostensen M, Grutzkau A, Radbruch A, Burmester GR, Villiger PM. Reactivation of rheumatoid arthritis after pregnancy: increased phagocyte and recurring lymphocyte gene activity. Arthritis Rheum. 2008 Oct;58(10):2981-92. doi: 10.1002/art.23907. PMID 18821679
- [Background] Jedel S, Hoffman A, Merriman P, Swanson B, Voigt R, Rajan KB, Shaikh M, Li H, Keshavarzian A. A randomized controlled trial of mindfulness-based stress reduction to prevent flare-up in patients with inactive ulcerative colitis. Digestion. 2014;89(2):142-55. doi: 10.1159/000356316. Epub 2014 Feb 14. PMID 24557009
- [Background] Kalanthroff E, Henik A, Derakshan N, Usher M. Anxiety, emotional distraction, and attentional control in the Stroop task. Emotion. 2016 Apr;16(3):293-300. doi: 10.1037/emo0000129. Epub 2015 Nov 16. PMID 26571078
- [Background] Kane HS, Dunkel Schetter C, Glynn LM, Hobel CJ, Sandman CA. Pregnancy anxiety and prenatal cortisol trajectories. Biol Psychol. 2014 Jul;100:13-9. doi: 10.1016/j.biopsycho.2014.04.003. Epub 2014 Apr 21. PMID 24769094
- [Background] 49. Kasper, S., den Boer, J.A., Ad Sitsen, J.M., 2003. Handbook of Depression and Anxiety: A Biological Approach, 2nd Ed. Marcel Dekker Inc., New York.
- [Background] Kim C, Brawarsky P, Jackson RA, Fuentes-Afflick E, Haas JS. Changes in health status experienced by women with gestational diabetes and pregnancy-induced hypertensive disorders. J Womens Health (Larchmt). 2005 Oct;14(8):729-36. doi: 10.1089/jwh.2005.14.729. PMID 16232105
- [Background] Kivlighan KT, DiPietro JA, Costigan KA, Laudenslager ML. Diurnal rhythm of cortisol during late pregnancy: associations with maternal psychological well-being and fetal growth. Psychoneuroendocrinology. 2008 Oct;33(9):1225-35. doi: 10.1016/j.psyneuen.2008.06.008. Epub 2008 Aug 8. PMID 18692319
- [Background] Kurki T, Hiilesmaa V, Raitasalo R, Mattila H, Ylikorkala O. Depression and anxiety in early pregnancy and risk for preeclampsia. Obstet Gynecol. 2000 Apr;95(4):487-90. doi: 10.1016/s0029-7844(99)00602-x. PMID 10725477
- [Background] Lambert JJ, Belelli D, Hill-Venning C, Peters JA. Neurosteroids and GABAA receptor function. Trends Pharmacol Sci. 1995 Sep;16(9):295-303. doi: 10.1016/s0165-6147(00)89058-6. PMID 7482994
- [Background] Maes M, Bosmans E, Ombelet W. In the puerperium, primiparae exhibit higher levels of anxiety and serum peptidase activity and greater immune responses than multiparae. J Clin Psychiatry. 2004 Jan;65(1):71-6. doi: 10.4088/jcp.v65n0112. PMID 14744172
- [Background] Maes M, Lin AH, Ombelet W, Stevens K, Kenis G, De Jongh R, Cox J, Bosmans E. Immune activation in the early puerperium is related to postpartum anxiety and depressive symptoms. Psychoneuroendocrinology. 2000 Feb;25(2):121-37. doi: 10.1016/s0306-4530(99)00043-8. PMID 10674277
- [Background] Maes M, Song C, Lin A, De Jongh R, Van Gastel A, Kenis G, Bosmans E, De Meester I, Benoy I, Neels H, Demedts P, Janca A, Scharpe S, Smith RS. The effects of psychological stress on humans: increased production of pro-inflammatory cytokines and a Th1-like response in stress-induced anxiety. Cytokine. 1998 Apr;10(4):313-8. doi: 10.1006/cyto.1997.0290. PMID 9617578
- [Background] Maes M, Verkerk R, Bonaccorso S, Ombelet W, Bosmans E, Scharpe S. Depressive and anxiety symptoms in the early puerperium are related to increased degradation of tryptophan into kynurenine, a phenomenon which is related to immune activation. Life Sci. 2002 Sep 6;71(16):1837-48. doi: 10.1016/s0024-3205(02)01853-2. PMID 12175700
- [Background] Makhseed M, Raghupathy R, Azizieh F, Farhat R, Hassan N, Bandar A. Circulating cytokines and CD30 in normal human pregnancy and recurrent spontaneous abortions. Hum Reprod. 2000 Sep;15(9):2011-7. doi: 10.1093/humrep/15.9.2011. PMID 10967006
- [Background] Matthey S, Barnett B, Howie P, Kavanagh DJ. Diagnosing postpartum depression in mothers and fathers: whatever happened to anxiety? J Affect Disord. 2003 Apr;74(2):139-47. doi: 10.1016/s0165-0327(02)00012-5. PMID 12706515
- [Background] Mautner E, Greimel E, Trutnovsky G, Daghofer F, Egger JW, Lang U. Quality of life outcomes in pregnancy and postpartum complicated by hypertensive disorders, gestational diabetes, and preterm birth. J Psychosom Obstet Gynaecol. 2009 Dec;30(4):231-7. doi: 10.3109/01674820903254757. PMID 19845493
- [Background] Mendelson T, DiPietro JA, Costigan KA, Chen P, Henderson JL. Associations of maternal psychological factors with umbilical and uterine blood flow. J Psychosom Obstet Gynaecol. 2011 Mar;32(1):3-9. doi: 10.3109/0167482X.2010.544427. Epub 2011 Jan 10. PMID 21219117
- [Background] Miaskowski C, Elboim C, Paul SM, Mastick J, Cooper BA, Levine JD, Aouizerat BE. Polymorphisms in Tumor Necrosis Factor-alpha Are Associated With Higher Anxiety Levels in Women After Breast Cancer Surgery. Clin Breast Cancer. 2016 Feb;16(1):63-71.e3. doi: 10.1016/j.clbc.2014.12.001. Epub 2014 Dec 24. PMID 25813148
- [Background] Milgrom J, Gemmill AW, Bilszta JL, Hayes B, Barnett B, Brooks J, Ericksen J, Ellwood D, Buist A. Antenatal risk factors for postnatal depression: a large prospective study. J Affect Disord. 2008 May;108(1-2):147-57. doi: 10.1016/j.jad.2007.10.014. Epub 2007 Dec 18. PMID 18067974
- [Background] O'Connor TG, Tang W, Gilchrist MA, Moynihan JA, Pressman EK, Blackmore ER. Diurnal cortisol patterns and psychiatric symptoms in pregnancy: short-term longitudinal study. Biol Psychol. 2014 Feb;96:35-41. doi: 10.1016/j.biopsycho.2013.11.002. Epub 2013 Nov 12. PMID 24239618
- [Background] O'Donnell KJ, Bugge Jensen A, Freeman L, Khalife N, O'Connor TG, Glover V. Maternal prenatal anxiety and downregulation of placental 11beta-HSD2. Psychoneuroendocrinology. 2012 Jun;37(6):818-26. doi: 10.1016/j.psyneuen.2011.09.014. Epub 2011 Oct 15. PMID 22001010
- [Background] Oglodek EA, Szota AM, Just MJ, Mos DM, Araszkiewicz A. The MCP-1, CCL-5 and SDF-1 chemokines as pro-inflammatory markers in generalized anxiety disorder and personality disorders. Pharmacol Rep. 2015 Feb;67(1):85-9. doi: 10.1016/j.pharep.2014.08.006. Epub 2014 Aug 21. PMID 25560580
- [Background] Oliveira Miranda D, Soares de Lima TA, Ribeiro Azevedo L, Feres O, Ribeiro da Rocha JJ, Pereira-da-Silva G. Proinflammatory cytokines correlate with depression and anxiety in colorectal cancer patients. Biomed Res Int. 2014;2014:739650. doi: 10.1155/2014/739650. Epub 2014 Sep 17. PMID 25309921
- [Background] Orr ST, James SA, Blackmore Prince C. Maternal prenatal depressive symptoms and spontaneous preterm births among African-American women in Baltimore, Maryland. Am J Epidemiol. 2002 Nov 1;156(9):797-802. doi: 10.1093/aje/kwf131. PMID 12396996
- [Background] Osborne L, Clive M, Kimmel M, Gispen F, Guintivano J, Brown T, Cox O, Judy J, Meilman S, Braier A, Beckmann MW, Kornhuber J, Fasching PA, Goes F, Payne JL, Binder EB, Kaminsky Z. Replication of Epigenetic Postpartum Depression Biomarkers and Variation with Hormone Levels. Neuropsychopharmacology. 2016 May;41(6):1648-58. doi: 10.1038/npp.2015.333. Epub 2015 Oct 27. PMID 26503311
- [Background] Osborne LM, Monk C. Perinatal depression--the fourth inflammatory morbidity of pregnancy?: Theory and literature review. Psychoneuroendocrinology. 2013 Oct;38(10):1929-52. doi: 10.1016/j.psyneuen.2013.03.019. Epub 2013 Apr 20. PMID 23608136
- [Background] Palmsten K, Setoguchi S, Margulis AV, Patrick AR, Hernandez-Diaz S. Elevated risk of preeclampsia in pregnant women with depression: depression or antidepressants? Am J Epidemiol. 2012 May 15;175(10):988-97. doi: 10.1093/aje/kwr394. Epub 2012 Mar 22. PMID 22442287
- [Background] Pan W. Akaike's information criterion in generalized estimating equations. Biometrics. 2001 Mar;57(1):120-5. doi: 10.1111/j.0006-341x.2001.00120.x. PMID 11252586
- [Background] Patchev VK, Hassan AH, Holsboer DF, Almeida OF. The neurosteroid tetrahydroprogesterone attenuates the endocrine response to stress and exerts glucocorticoid-like effects on vasopressin gene transcription in the rat hypothalamus. Neuropsychopharmacology. 1996 Dec;15(6):533-40. doi: 10.1016/S0893-133X(96)00096-6. PMID 8946427
- [Background] Phillips J, Sharpe L, Matthey S. Rates of depressive and anxiety disorders in a residential mother-infant unit for unsettled infants. Aust N Z J Psychiatry. 2007 Oct;41(10):836-42. doi: 10.1080/00048670701579108. PMID 17828657
- [Background] Phillips J, Sharpe L, Matthey S, Charles M. Maternally focused worry. Arch Womens Ment Health. 2009 Dec;12(6):409-18. doi: 10.1007/s00737-009-0091-4. Epub 2009 Jul 21. PMID 19626414
- [Background] Raghupathy R, Al-Azemi M. Modulation of Cytokine Production by the Dydrogesterone Metabolite Dihydrodydrogesterone. Am J Reprod Immunol. 2015 Nov;74(5):419-26. doi: 10.1111/aji.12418. Epub 2015 Aug 7. PMID 26250154
- [Background] Robinson DP, Klein SL. Pregnancy and pregnancy-associated hormones alter immune responses and disease pathogenesis. Horm Behav. 2012 Aug;62(3):263-71. doi: 10.1016/j.yhbeh.2012.02.023. Epub 2012 Mar 3. PMID 22406114
- [Background] Rosenkranz MA, Davidson RJ, Maccoon DG, Sheridan JF, Kalin NH, Lutz A. A comparison of mindfulness-based stress reduction and an active control in modulation of neurogenic inflammation. Brain Behav Immun. 2013 Jan;27(1):174-84. doi: 10.1016/j.bbi.2012.10.013. Epub 2012 Oct 22. PMID 23092711
- [Background] Ross LE, McLean LM. Anxiety disorders during pregnancy and the postpartum period: A systematic review. J Clin Psychiatry. 2006 Aug;67(8):1285-98. doi: 10.4088/jcp.v67n0818. PMID 16965210
- [Background] Russell EJ, Fawcett JM, Mazmanian D. Risk of obsessive-compulsive disorder in pregnant and postpartum women: a meta-analysis. J Clin Psychiatry. 2013 Apr;74(4):377-85. doi: 10.4088/JCP.12r07917. PMID 23656845
- [Background] Schofield CA, Battle CL, Howard M, Ortiz-Hernandez S. Symptoms of the anxiety disorders in a perinatal psychiatric sample: a chart review. J Nerv Ment Dis. 2014 Feb;202(2):154-60. doi: 10.1097/NMD.0000000000000086. PMID 24469528
- [Background] Schumacher M, Mattern C, Ghoumari A, Oudinet JP, Liere P, Labombarda F, Sitruk-Ware R, De Nicola AF, Guennoun R. Revisiting the roles of progesterone and allopregnanolone in the nervous system: resurgence of the progesterone receptors. Prog Neurobiol. 2014 Feb;113:6-39. doi: 10.1016/j.pneurobio.2013.09.004. Epub 2013 Oct 27. PMID 24172649
- [Background] 72. Segal ZV, Williams JM, Teasdale JD (2002) Mindfulness-based cognitive therapy for depression. Guilford, New York
- [Background] 73. Segal ZV, Williams JM, Teasdale JD (2013) Mindfulness-based cognitive therapy for depression second edition. Guilford, New York
- [Background] Shadigian E, Bauer ST. Pregnancy-associated death: a qualitative systematic review of homicide and suicide. Obstet Gynecol Surv. 2005 Mar;60(3):183-90. doi: 10.1097/01.ogx.0000155967.72418.6b. PMID 16570396
- [Background] Slattery MJ, Dubbert BK, Allen AJ, Leonard HL, Swedo SE, Gourley MF. Prevalence of obsessive-compulsive disorder in patients with systemic lupus erythematosus. J Clin Psychiatry. 2004 Mar;65(3):301-6. doi: 10.4088/jcp.v65n0303. PMID 15096067
- [Background] Sutter-Dallay AL, Giaconne-Marcesche V, Glatigny-Dallay E, Verdoux H. Women with anxiety disorders during pregnancy are at increased risk of intense postnatal depressive symptoms: a prospective survey of the MATQUID cohort. Eur Psychiatry. 2004 Dec;19(8):459-63. doi: 10.1016/j.eurpsy.2004.09.025. PMID 15589703
- [Background] Tamasi L, Horvath I, Bohacs A, Muller V, Losonczy G, Schatz M. Asthma in pregnancy--immunological changes and clinical management. Respir Med. 2011 Feb;105(2):159-64. doi: 10.1016/j.rmed.2010.11.006. Epub 2010 Dec 8. PMID 21145223
- [Background] Vogelzangs N, Beekman AT, de Jonge P, Penninx BW. Anxiety disorders and inflammation in a large adult cohort. Transl Psychiatry. 2013 Apr 23;3(4):e249. doi: 10.1038/tp.2013.27. PMID 23612048
- [Background] Wohleb ES, Patterson JM, Sharma V, Quan N, Godbout JP, Sheridan JF. Knockdown of interleukin-1 receptor type-1 on endothelial cells attenuated stress-induced neuroinflammation and prevented anxiety-like behavior. J Neurosci. 2014 Feb 12;34(7):2583-91. doi: 10.1523/JNEUROSCI.3723-13.2014. PMID 24523548
- [Background] Zernicke KA, Campbell TS, Blustein PK, Fung TS, Johnson JA, Bacon SL, Carlson LE. Mindfulness-based stress reduction for the treatment of irritable bowel syndrome symptoms: a randomized wait-list controlled trial. Int J Behav Med. 2013 Sep;20(3):385-96. doi: 10.1007/s12529-012-9241-6. PMID 22618308
- [Derived] Riddle JN, Jager LR, Sherer M, Pangtey M, Osborne LM. Anxiety in pregnancy and stress responsiveness: An exploratory study of heart rate variability, cortisol, and alpha-amylase in the third trimester. J Neuroendocrinol. 2023 Jul;35(7):e13238. doi: 10.1111/jne.13238. Epub 2023 Mar 3. PMID 36866835
- See also: Hintze, J. PASS 12. 2013. NCSS, LLC. Kaysville, Utah, USA — http://www.ncss.com.